CLINICAL TRIAL: NCT03036982
Title: Remote Use of the Asthma Control Test (ACT) to Improve Care of Children With Asthma
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Andrew MacGinnitie, Associate Clinical Director, Division of Immunology, Boston Children's Hospital
Other Study IDs: FP01013808
Record Dates: First submitted 2015-07-27; First posted 2017-01-31 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Use of Mobile ACT: Will answer ACT (or cACT) and other asthma questions using mobile app

SUMMARY:
This study will assess whether adaption of the Asthma Control Test (ACT) and childhood Asthma Control Test (cACT) for mobile devices improves rate of completion and improves control of asthma in children and adolescents

DETAILED DESCRIPTION:
Asthma is the most prevalent chronic disease of childhood with an overall prevalence of 10%. While effective therapies exist to control symptoms and prevent exacerbations, many asthma patients experience significant morbidity including limitations on daily activities as well as asthma exacerbations that lead to missed school (and work for care givers) and necessitate emergency department visits and hospitalizations. Among children from lower socioeconomic statues and in black and Hispanic families, asthma incidence and severity are even greater. Reasons for this disparity included decreased access to effective asthma care, increased exposure to tobacco smoke and environmental allergens, and underutilization of controller medicines. These groups have significantly increased resource utilization due to emergency department visits and hospitalizations. Optimal care for asthma patients, especially those with at highest risk, will therefore require new strategies for evaluating ongoing control and providing direct feedback to patients.

We propose to transform the way asthma care is provided through the use of an innovative patient centered technology -Trivox Asthma - to improve quality of care and outcomes for asthma patients while reducing the cost of care. Specifically we will extend Trivox Health to facilitate closer monitoring of patients with asthma through the existing web platform and a new mobile interface. This will allow asthma patients, their parents and school nurses to remotely input data on asthma control through smartphones and/or tablets. We will use the ACT+, an expansion of a validated measure currently utilized in both primary care and specialty clinics, to measure both asthma control and risk.

Effectiveness of this intervention will be measured by examining resource utilization and ongoing asthma control.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma
* Cared for at Boston Children's Hospital (Primary or secondary care)

Exclusion Criteria:

* Age <4 or >21

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with asthma seen in one of the clinics caring for patients with asthma at Boston Children's Hospital Age 4-21
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Well-controlled asthma | Each month for one calendar year
  Percent of ACT scores with value of 20 or greater

SECONDARY OUTCOMES:
Asthma Emergency Department visits and hospitalizations | Total Emergency Department Visits and hospitalizations with asthma as one of top diagnosis in one year
  Asked every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew MacGinnitie, MD PhD, Principal Investigator — Boston Children's Hosptial
Locations (1):
- Boston Childrens Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Will make deidentified data available for other researchers